CLINICAL TRIAL: NCT05934487
Title: A Prospective, Multi-Center, Open Label, Randomized Control Clinical Trial Evaluating the Safety and Efficacy of the Cordella™ Pulmonary Artery Sensor System in New York Heart Association (NYHA) Class II-III Heart Failure Patients
Brief Title: PROACTIVE-HF-2 Trial Heart Failure NYHA Class II and III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ETX-HFS-PA-04
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure
Keywords: Heart Failure; Heart Disease; Cardiovascular Disease; Pulmonary Artery Pressure
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- NYHA II Treatment Arm (Experimental): All subjects will receive the Cordella Sensor.
  Clinicians will manage the subjects to target PAP per protocols specific Treatment Guidelines and according to Guideline-Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA II Active Control Arm (Experimental): All subjects will receive the Cordella Sensor.
  Clinicians will manage subjects using the subjects daily data trends (BP, weight, HR, SpO2 symptoms) according to Guideline Directed Medical Therapy. Once the primary endpoint (24 months) is met, subjects and clinicians will be unblinded to PAP.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA II Crossover Arm (Experimental): All subjects will receive the Cordella Sensor.
  At least 12 months following implant and following an adjudicated HFH, subjects in the Active Control Arm can qualify to crossover to the Crossover Arm and both patients and clinicians would then be unmasked to PAP. Clinicians will then manage the subjects to target PAP per protocols specific Treatment Guidelines and according to Guideline-Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA III Phase I Treatment Arm (Experimental): All subjects will receive the Cordella Sensor.
  Clinicians will manage the subjects to target PAP per protocols specific Treatment Guidelines and according to Guideline-Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA III Phase I Active Control Arm (Experimental): All subjects will receive the Cordella Sensor.
  Clinicians will manage subjects using the subjects daily data trends (BP, weight, HR, SpO2 symptoms) according to Guideline Directed Medical Therapy. Once the primary endpoint (6 months) is met, subjects and clinicians will be unblinded to PAP.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA III Clinician-Directed Patient Self-Management Arm (randomized) (Experimental): This is Phase II / Randomization #2 following implant provided patient meets eligiibity criteria.
  Subjects will be instructed to take their PAP measurements daily in addition to their weight, BP, SpO2, and HR. All data, including PAP, will be visible to the patient. Subjects will manage their diuretics per protocol specific Clinician-Directed Patient Self-Management Treatment Guidelines. Clinicians will oversee the patient self-management to target PAP per protocol specific Treatment Guidelines and according to Guideline-Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA III Clinician Management Arm (randomized) (Experimental): This is Phase II / Randomization #2 following implant provided patient meets eligiibity criteria.
  Subjects will be instructed to take their PAP measurements daily in addition to their weight, BP, SpO2, and HR. All data, including PAP, will be visible to the patient. Subjects will manage their diuretics per protocol specific Clinician-Directed Patient Self-Management Treatment Guidelines. Clinicians will manage the patients to target PAP per protocols specific to Treatment Guidelines and according to Guideline Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System
- NYHA III Clinician Management Arm (Not randomized) (Experimental): Subject will not be randomized if they do not meet eligibility criteria to potentially be randomized to Clinician-Directed Patient Self-Management.
  Subjects will be instructed to take their PAP measurements daily in addition to their weight, BP, SpO2, and HR. All data, including PAP, will be visible to the patient. Subjects will manage their diuretics per protocol specific Clinician-Directed Patient Self-Management Treatment Guidelines. Clinicians will manage the patients to target PAP per protocols specific to Treatment Guidelines and according to Guideline Directed Medical Therapy.
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System

INTERVENTIONS:
Device: Cordella™ Pulmonary Artery Sensor System — The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management, with the goal of reducing heart failure hospitalizations. The system comprises of seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  Cordella Sensor Cordella Delivery System myCordella Patient Reader Reader Dock Cordella Calibration Equipment (CalEQ) myCordella Tablet Cordella Data Analysis Platform (CDAP)

SUMMARY:
This is a prospective, multi-center, open label, randomized control clinical trial evaluating the safety and efficacy of the Cordella™ Pulmonary Artery Sensor System in NYHA Class II-III Heart Failure Patients (PROACTIVE-HF-2 Trial).

The study contains of 5 arms:

NYHA II Cohort - To demonstrate safety and efficacy of the Cordella PA Sensor System in NYHA Class II HF patients, where patients have daily access to PAP data.

* Treatment Arm (Group 1)
* Active Control Arm (Group 2)
* Crossover Arm (Group 3)

NYHA III Cohort - To demonstrate safety and efficacy of the Cordella PA Sensor System in NYHA Class III HF patients, where patients have daily access to PAP data, including a randomized sub-study to evaluate a clinician-directed patient self-management strategy.

ELIGIBILITY:
Inclusion Criteria 1. Subject has given written informed consent 2. Male or female, at least 18 years of age 3. Diagnosis and treatment of HF (regardless of LVEF) for ≥ 3 months and NYHA Class II HF (NYHA II Cohort) or NYHA III (NYHA III Cohort) at time of Screening

4. Subjects should be receiving appropriate medical therapy for heart failure according to current AHA/ACC guidelines as standard-of-care for HF therapy in the United States, or current ESC guidelines for HF treatment in Europe for at least 30 days prior to the Screening/Enrollment visit. Stable is defined as no more than a 100% increase or 50% decrease in dose. These criteria may be waived if a subject is intolerant of ACE-I, ARB, ARNI), MRA, beta-blockers, or SGLT2i, subject is unable to afford these agents, subject has contraindications to these agents, or these agents are not indicated under the Guidelines. Such intolerance, lack of affordability, contraindications, or lack of indications must be documented.

1. HFrEF (EF < 50%): Subject has been on stable medications maximized to the subject's tolerance of ACE-I or ARB or ARNI, MRA, beta-blockers, and SGLT2i as determined by the study investigator for at least 30 days prior to Screening/Enrollment
2. HFpEF (EF ≥ 50%): Subject has been on stable medication maximized to the subject's tolerance of SGLT2i as determined by the study investigator for at least 30 days prior to Screening/Enrollment 5. NYHA II Cohort- HF related hospitalization within 6 months (last hospitalization should be 30 days before Screening /Enrollment) 5. NYHA III Cohort -HF related hospitalization within 12 month (last hospitalization should be 30 days before Screening/Enrollment)

   6. Subjects should be on diuretic therapy (≥40 mg] furosemide or equivalent) for ≥ 1 month at time of Screening

   7. Subjects who are physically able to hold the myCordella™ Patient Reader unit (approximate weight 1.3lb) against the ventral thoracic surface for up to 2 minutes per day while in a seated position, as well as dock and undock the myCordella™ Patient Reader

   8. Subjects with sufficient eyesight, hearing, and mental capacity to respond to the myCordella™ Patient Reader's audio/visual cues and operate the myCordella™ Patient Reader

   9. Subject has sufficient Cellular and/ or Wi- Fi Internet coverage at home

   10. Subject agrees to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up

   Exclusion Criteria:
   1. ACC/AHA Stage D refractory HF (including a known history of >24 hours of IV inotropic therapy to support circulation within the past 6 months (other than relation to a procedure))
   2. Subjects with history of recurrent pulmonary embolism (≥2 episodes within 5 years prior to Screening Visit) and/or deep vein thrombosis in the femoral or IJ vein used for access (< 3 month prior to Screening Visit)
   3. Subjects with a resting systolic blood pressure <90 mmHg and/ or severe pre-capillary pulmonary hypertension with a pulmonary artery systolic pressure of ≥70 mm/Hg with pulmonary capillary wedge pressure ≤ 15 mmHg at the Cordella PA Sensor Implant RHC (V2)
   4. Subjects who have had a major cardiovascular (CV) event (e.g., myocardial infarction, stroke) within 3 months of the Screening Visit
   5. Unrepaired severe valvular disease
   6. Subjects with significant congenital heart disease that has not been repaired and would prevent implantation of the Cordella PA Sensor or mechanical/tissue right heart valve(s)
   7. Subjects with known coagulation disorders
   8. Subjects with a hypersensitivity or allergy to platelet aggregation inhibitors including aspirin, clopidogrel, prasugrel, and ticagrelor; or patients unable to take dual antiplatelet or anticoagulants for one-month post implant
   9. Known history of life-threatening allergy to contrast dye.
   10. Subjects whereby RHC is contraindicated
   11. Subjects with an active infection at the Cordella Sensor Implant Visit
   12. Subjects with a GFR <20 ml/min or who are on chronic renal dialysis
   13. Implanted with Cardiac Resynchronization Therapy-Pacemaker (CRT-P) or Cardiac Resynchronization Therapy-Defibrillator (CRT-D), or having undergone mitral/tricuspid valve repair/replacement within 90 days or catheter ablation for atrial fibrillation within 30 days prior to screening visit
   14. Received or are likely to receive an advanced therapy (e.g., durable mechanical circulatory support or lung or heart transplant) in the next 24 months
   15. Subjects who are pregnant or breastfeeding
   16. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
   17. Severe illness, other than heart disease, which would limit survival to <2 years
   18. Subjects whose clinical condition, in the opinion of the Investigator, makes them an unsuitable candidate for the study
   19. Subjects enrolled in another investigational trial with an active Treatment Arm
   20. Subject who is in custody by order of an authority or a court of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy- NYHA II Cohort - A composite of first HF event or death from Cardiovascular Death up to 24 months. | 24 months
  A composite endpoint of first HF event or death from CVD up to 24 months.
Efficacy- NYHA III Cohort (Phase I) - a composite of HF events or death from cardiovascular disease at 6 months | 12 months
  A composite of HF events or death from cardiovascular disease at 6 months
Safety- Randomized Arm- Freedom from device/system related complication | 24 months
  Freedom from device/system related complication at 24 months
Safety- Randomized Arm-Freedom from pressure sensor failure | 24 months
  Freedom from pressure sensor failure at 24 months
Safety- Single Arm-Freedom from device/system related complication | 12 months
  Freedom from device/system related complication at 12 months
Safety- Single Arm- Freedom from pressure sensor failure | 12 months
  Freedom from pressure sensor failure at 12 months
Efficacy- NYHA III Cohort (Phase II) - A test of non-inferiority at 12 months of the percentage of patients at or below trend seated mPAP of 25 mmHg in (i) Clinician-Directed Patient Self-Management vs. (ii) Clinician Management Arm | 12 months
  A test of non-inferiority at 12 months of the percentage of patients at or below trend seated mPAP of 25 mmHg in (i) Clinician-Directed Patient Self-Management vs. (ii) Clinician Management Arm

SECONDARY OUTCOMES:
Efficacy - NYHA II Cohort & NYHA III Cohort - HF Hospitalizations | 12 months, 18 months and 24 months
  -Incidence of HFH at 12, 18, and 24 months
Efficacy - NYHA II Cohort & NYHA III Cohort- HF Hospitalizations | 12 months and 24 months
  -Number of HFH at 12- and 24-months post-implant compared to the number of HFH in the 12 and 24 months prior to implant
Efficacy - NYHA II Cohort & NYHA III Cohort - HF Hospitalizations | 12 month
  Combined outcome of :
  1. First and recurrent HF Hospitalizations
  2. Urgent HF Visits
  3. all-cause mortality
Efficacy - NYHA II Cohort & NYHA III Cohort - HF Hospitalizations | Duration of study (to 5 years)
  Length of stay
Efficacy - NYHA II Cohort & NYHA III Cohort - All-cause mortality | Duration of study (to 5 years)
  All-cause mortality
Efficacy - NYHA II Cohort & NYHA III Cohort - Death from cardiovascular disease | Duration of study (to 5 years)
  Death from cardiovascular disease
Efficacy - NYHA II Cohort & NYHA III Cohort - Urgent HF visits | Duration of study (to 5 years)
  Urgent HF visits
Efficacy - NYHA II Cohort - Incidence of HF hospitalizations or all-cause mortality | 12 months
  Incidence of HF hospitalizations or all-cause mortality
Efficacy - NYHA III Cohort - Composite of first HF event (HF hospitalization or urgent HF visit or death from cardiovascular disease (CVD) | Up to 24 months
  Composite of first HF event (HF hospitalization or urgent HF visit or
Eff-NYHA II Cohort & NYHA III Cohort -time to death, # HFH or urgent HF visits, time to first HFH or urgent HF visit, diff >/= 15 KCCQ BSL to 24 mos,diff >/= 10 in KCCQ BSL to 24 mos, diff >/= 5 in KCCQ BSL to 24 mos, diff >/= 30m in 6 MWT BSL to 24 mos | Duration of study (to 5 years)
  -time to death, # HFH or urgent HF visits, time to first HFH or urgent HF visit, diff >/= 15 KCCQ BSL to 24 mos,diff >/= 10 in KCCQ BSL to 24 mos, diff >/= 5 in KCCQ BSL to 24 mos, diff >/= 30m in 6 MWT BSL to 24 mos
Efficacy - NYHA II Cohort & NYHA III Cohort - Various measurements via ECHO and evaluated by ECHO core lab at Baseline, 12, 24, 36, 48 and 60 months. | Duration of study (to 5 years)
  Various measurements via ECHO and evaluated by ECHO core lab at Baseline, 12, 24, 36, 48 and 60 months.
Efficacy - NYHA II Cohort & NYHA III Cohort - Heart failure related medication changes | Duration of study (to 5 years)
  Heart failure related medication changes
Efficacy - NYHA II Cohort & NYHA III Cohort - Change in PAP from baseline | Duration of study (to 5 years)
  Change in PAP from baseline
Efficacy - NYHA II Cohort & NYHA III Cohort - Change in PAP from baseline as measured by echocardiogram (ECHO) and evaluated by anECHO core lab at 12, 24, 36, 48, and 60 months | Duration of study (to 5 years)
  Change in PAP from baseline as measured by echocardiogram (ECHO) and evaluated by an ECHO core lab at 12, 24, 36, 48, and 60 months
Efficacy - NYHA II Cohort & NYHA III Cohort - Patient Outcome Measures as measured by KCCQ, Brief Illness Perception Questionnaire, andEuroQol-5 Dimensions-5 Level (EQ-5D-5L) | Duration of study (to 5 years)
  Patient Outcome Measures as measured by KCCQ, Brief Illness Perception Questionnaire, and EuroQol-5 Dimensions-5 Level (EQ-5D-5L)
Efficacy - NYHA II Cohort & NYHA III Cohort - Functional status improvement as measured by NYHA classification and 6MWT | Duration of study (to 5 years)
  Functional status improvement as measured by NYHA classification and 6MWT
Efficacy - NYHA II Cohort & NYHA III Cohort - HFH stratified by ejection fraction (HFrEF, HFmrEF, HFpEF, and HF recovered EF) and baselineenrollment ECHO estimated systolic PAP | Duration of study (to 5 years)
  HFH stratified by ejection fraction (HFrEF,
Efficacy - NYHA II Cohort & NYHA III Cohort - Mortality by baseline EF (HFrEF, HFmrEF, HFpEF, HF recovered EF), and baseline enrollmentECHO estimated systolic PAP | Duration of study (to 5 years)
  Mortality by baseline EF (HFrEF, HFmrEF,
Efficacy - NYHA II Cohort & NYHA III Cohort - Days alive outside hospital (DAOH) | Duration of study (to 5 years)
  Days alive outside hospital (DAOH)
Efficacy - NYHA II Cohort & NYHA III Cohort - Health Economic Analysis | Duration of study (to 5 years)
  Health Economic Analysis
Efficacy - NYHA II Cohort & NYHA III Cohort - Adherence to regular PAP and vital sign measurements including a sub-analysis on subjectswho move to another area of the country | Duration of study (to 5 years)
  Adherence to regular PAP and vital sign measurements including a sub-analysis on subjects who move to another area of the country
Safety - NYHA II Cohort - Freedom from device/system related complications at 12 months | Duration of study (to 5 years)
  Freedom from device/system related complications at 12 months
Safety - NYHA III Cohort - Freedom from pressure sensor failure at 12 months | Duration of study (to 5 years)
  Freedom from pressure sensor failure at 12 months
Safety - NYHA II Cohort & NYHA III Cohort - Pressure sensor failure rate throughout the study | Duration of study (to 5 years)
  Pressure sensor failure rate throughout the study
Safety - NYHA II Cohort & NYHA III Cohort - Frequency of serious adverse events throughout the study | Duration of study (to 5 years)
  Frequency of serious adverse events throughout the study
Safety - NYHA II Cohort & NYHA III Cohort - Frequency of implant procedure and procedure related adverse events and serious adverse events | Duration of study (to 5 years)
  Frequency of implant procedure and procedure related adverse events and serious adverse events
Safety - NYHA III Cohort - Freedom from device/system related complications at 24 months | Duration of study (to 5 years)
  Freedom from device/system related complications at 24 months
Safety - NYHA III Cohort - Freedom from pressure sensor failure at 24 months | Duration of study (to 5 years)
  Freedom from pressure sensor failure at 24 months

OTHER OUTCOMES:
Safety - NYHA III Cohort Phase II only: Incidence of serious adverse events at 12 months post Phase II randomization | 12 months
  Incidence of serious adverse events at 12 months post Phase II randomization

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sauerland, Study Director — Endotronix, Inc.
Locations (49):
- United States (46):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Baptist Health South Florida, Miami, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Piedmont, Atlanta, Georgia
  - Advocate Health System, Downers Grove, Illinois
  - Heart Care Centers of Illinois (HCCI), Palos Park, Illinois
  - Ascension St. Vincent's, Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - MedStar, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Ascension Providence Hospital Cardiology - Heart Cardiology, Howell, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Centra Care Heart Center, Saint Cloud, Minnesota
  - St. Lukes/ Mid-American Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Mount Sinai West, New York, New York
  - Mount Sinai, New York, New York
  - Lenox Hill/ Northwell Health, New York, New York
  - Stony Brook University Med Center, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - The Christ Hospital- Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospital (Cleveland), Cleveland, Ohio
  - Providence St. Vincent's - Portland, Portland, Oregon
  - Oregon Health Science Portland, Portland, Oregon
  - Penn State Health, Hershey, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - PRISMA Health- Upstate, Greenville, South Carolina
  - Sanford, Sioux Falls, South Dakota
  - Vanderbilt, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Medical City Healthcare Dallas, Dallas, Texas
  - Baylor Scott & White -Dallas, Fort Worth, Texas
  - Baylor/Texas Heart, Houston, Texas
  - Methodist San Antonio, San Antonio, Texas
  - Baylor - Temple, Temple, Texas
  - University of Vermont, Burlington, Vermont
  - Providence Everett, Everett, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Advocate Aurora St. Luke's, Milwaukee, Wisconsin
- Belgium (2):
  - AZORG Aalst, Aalst, Aalst
  - UZ Brussel, Brussels
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No